CLINICAL TRIAL: NCT01766700
Title: The Role of No-Calorie Sweetened Beverages Within a Weight Loss Behavior Change Program and During Subsequent Weight Maintenance
Brief Title: The Role of No-Calorie Beverages Within a Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12-1063
Record Dates: First submitted 2012-10-03; First posted 2013-01-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Obesity, weight loss, weight maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No calorie beverages (Experimental): 2 no calorie beverages per day.
  Interventions: Behavioral: 2 no calorie beverages per day
- Water (Active Comparator): 2 water beverages per day.
  Interventions: Behavioral: 2 water beverages per day

INTERVENTIONS:
Behavioral: 2 no calorie beverages per day — Weekly and monthly lifestyle weight loss/maintenance classes.
  Other Names: 2 non-nutritive sweetened beverages per day
  Arms: No calorie beverages
Behavioral: 2 water beverages per day — Weekly and monthly lifestyle weight loss/maintenance classes.
  Other Names: water only group
  Arms: Water

SUMMARY:
The no calorie drink study is looking for over 300 people to participate. The study is evaluating the effect of no calorie beverages on weight loss and weight maintained over time in people who drink diet beverages every day as compared to water only drinkers during the 1 year study period.

DETAILED DESCRIPTION:
This investigation aims to test the hypothesis that the amount of weight lost and maintained over time in an intensive behavioral weight management program will be equivalent in subjects consuming beverages containing no calorie sweeteners as compared to water beverages.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 27 - 40 kg/m2
* Must drink no calorie, sweetened drinks

Exclusion Criteria

* Cardiovascular disease
* Uncontrolled blood pressure
* Smoker
* Medications that affecting metabolism
* Oral steroids
* History of stroke or seizures
* Thyroid disease
* Type 1 or 2 diabetes
* Cushings syndrome
* Renal disease
* Liver disease
* Cancer in the past 5 years
* HIV
* Active tuberculosis
* Major psychiatric disorders

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
This investigation is an equivalency trial to determine whether weight loss differs between subjects consuming beverages containing no calorie sweeteners as compared to water drinkers at 12 weeks. | Data will be measured at 12 weeks.

SECONDARY OUTCOMES:
This investigation is an equivalency trial to determine whether weight lost and maintained during the 1 year study differs between subjects consuming beverages containing no calorie sweeteners as compared to water drinkers. | Data will be collected at end of study.

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, PhD, Principal Investigator — University of Colorado, Denver; Gary Foster, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Peters JC, Wyatt HR, Foster GD, Pan Z, Wojtanowski AC, Vander Veur SS, Herring SJ, Brill C, Hill JO. The effects of water and non-nutritive sweetened beverages on weight loss during a 12-week weight loss treatment program. Obesity (Silver Spring). 2014 Jun;22(6):1415-21. doi: 10.1002/oby.20737. PMID 24862170